CLINICAL TRIAL: NCT02834325
Title: Predicting Failure of High Flow Nasal Cannula in Pneumonia Patients With Hypoxemic Respiratory Failure: The Utility of ROX Index
Brief Title: Predicting Success of HFNC: The Utility of the ROX Index
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)101/2011
Record Dates: First submitted 2015-08-31; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Acute Respiratory Failure; Pneumonia
Keywords: high flow nasal cannula; success; failure; ROX index
MeSH Terms: conditions — Pneumonia | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- exit: HFNC with no need for mechanical ventilation
- failure: HFNC with need for mechanical ventilation
  Interventions: Procedure: mechanical ventilation

INTERVENTIONS:
Procedure: mechanical ventilation
  Groups: failure

SUMMARY:
The purpose of the study was to describe early predictors and to develop a prediction tool that accurately identifies the need for mechanical ventilation in pneumonia patients with acute respiratory failure treated with High Flow nasal cannula.

DETAILED DESCRIPTION:
Purpose The purpose of the study is to describe early predictors and to develop a prediction tool that accurately identifies the need for mechanical ventilation (MV) in pneumonia patients with hypoxemic acute respiratory failure (ARF) treated with high-flow nasal cannula (HFNC).

Materials and methods This is a 4-year prospective observational 2-center cohort study including patients with severe pneumonia treated with HFNC. High-flow nasal cannula failure was defined as need for MV. ROX index was defined as the ratio of pulse oximetry/fraction of inspired oxygen to respiratory rate.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute respiratory failure secondary to pneumonia receiving HFNC therapy

Exclusion Criteria:

* younger than 18 years old
* indication for mechanical ventilation at ICU admission
* limitation of therapeutic effort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute respiratory failure admitted to intensive care unit receiving high-flow nasal cannula treatment.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
prediction of need for mechanical ventilation using ROX index | through study completion, an average of 1 year
  participants will be followed during their stay in the ICU registering the days with HFNC treatment and their need or not for mechanical ventilation.

IPD SHARING:
Plan to Share IPD: No